CLINICAL TRIAL: NCT05910138
Title: Evaluation of Serum Levels of Interlukin-15 and Interlukin-21 in Patients With Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Samir George, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-06-05MS
Record Dates: First submitted 2023-06-11; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Active Comparator)
  Interventions: Diagnostic Test: Serum Interlukin-15; Diagnostic Test: Serum Interlukin-21
- control (Active Comparator)
  Interventions: Diagnostic Test: Serum Interlukin-15; Diagnostic Test: Serum Interlukin-21

INTERVENTIONS:
Diagnostic Test: Serum Interlukin-15 — Evaluate its serum level and detect its relation to the activity and severity of Alopecia Areata.
Diagnostic Test: Serum Interlukin-21 — Evaluate its serum level and detect its relation to the activity and severity of Alopecia Areata.

SUMMARY:
Alopecia areata (AA) is a type of non-cicatricial alopecia. The most common presentation of AA is localized patches of hair loss on the scalp. The extensive forms of AA presented as diffuse hair loss of the scalp (alopecia totalis) and diffuse hair loss through the entire body including the eyelashes and eyebrows (alopecia universalis).

AA affects approximately 2% of the general population. AA occurs at any age. The peak of incidence is higher in the second and third decades of life.

AA may be associated with several autoimmune diseases including thyroid diseases, lupus erythematosus, vitiligo, psoriasis, rheumatoid arthritis and inflammatory bowel disease. The frequency of the disease varies between geographically separate populations. These diseases associations suggest a relationship between AA and autoimmunity.

Human hair has an important cosmetic and communicational role. We may find significant psychological distress in persons with partial and complete hair loss. AA is associated with psychiatric morbidity especially anxiety and depression.

The pathogenesis of AA involves a complex interaction between genetic, environmental and immune factors. The histopathology of the disease differs according to the stage of the disease. In the acute stage of AA, there is a dense accumulation of lymphocytes (CD4 &CD8) around hair bulbs so called swarm of bees. In chronic stage, the inflammation may or may not resolve, but there is increase in number of catagen and, or telogen hair and pigmentary incontinence. In the recovery stage, there is minimal inflammation and increase in anagen hair.

T-helper17 cells are unique subset of T-helper cells which produce many interleukins (IL) e.g. IL-17A, IL-17F, IL-21, IL-22, IL-6 and tumor necrosis factor (TNF). The maturation of Th-17 needs the stimulation of naïve T cells by both TGF and IL-21. IL-21 is a cytokine that is produced mostly by activated CD4 T cells. It controls the differentiation and activity of T cells, B cells and NK cells. IL-21 could be a promising marker in the diagnosis of AA and also can be used as a marker of its activity.

IL-15 is a pleotropic cytokine that has multiple effects on different body cell types. It affects the function of cells of both innate and adaptive immune system. IL-15 is well known to promote lymphocytic development and suggested to play a role in some autoimmune diseases e.g. multiple sclerosis, rheumatoid arthritis, ulcerative colitis and celiac disease. IL-15 inhibits the well-known self-tolerance that mediated by activation - induced cell death, promotes maintenance of CD8+ memory T cells with induction of some cytokines which involved in autoimmune process e.g. TNF- and IL-1B. IL-15 is positively correlated with the number and the extent of AA so it could be a possible marker of AA severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex with active and stable AA.

Exclusion Criteria:

* -Pregnant patients.
* Lactating patients.
* Patients with other differential diagnoses of AA (Trichotillomania, temporal triangular alopecia, and tinea capitis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Serum levels of Interlukin-15 | 12 months
  Detection of its relation to activity and severity of Alopecia Areata
Evaluation of Serum levels of Interlukin-21 | 12 months
  Detection of its relation to activity and severity of Alopecia Areata

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Atwa MA, Youssef N, Bayoumy NM. T-helper 17 cytokines (interleukins 17, 21, 22, and 6, and tumor necrosis factor-alpha) in patients with alopecia areata: association with clinical type and severity. Int J Dermatol. 2016 Jun;55(6):666-72. doi: 10.1111/ijd.12808. Epub 2015 Jul 31. PMID 26235375
- [Background] Chaitra V, Rajalakshmi T, Kavdia R. Histopathologic profile of alopecia areata in Indian patients. Int J Trichology. 2010 Jan;2(1):14-7. doi: 10.4103/0974-7753.66906. PMID 21188017
- [Background] Darwin E, Hirt PA, Fertig R, Doliner B, Delcanto G, Jimenez JJ. Alopecia Areata: Review of Epidemiology, Clinical Features, Pathogenesis, and New Treatment Options. Int J Trichology. 2018 Mar-Apr;10(2):51-60. doi: 10.4103/ijt.ijt_99_17. PMID 29769777
- [Background] Ebrahim AA, Salem RM, El Fallah AA, Younis ET. Serum Interleukin-15 is a Marker of Alopecia Areata Severity. Int J Trichology. 2019 Jan-Feb;11(1):26-30. doi: 10.4103/ijt.ijt_80_18. PMID 30820130